CLINICAL TRIAL: NCT02398721
Title: A Prospective Randomized Study on Health-related Quality of Life of Patients With Incidental Small (<2cm) Asymptomatic Thyroid Nodules and Cost-effectiveness Analysis in Managing Small Incidental Thyroid Nodules
Brief Title: Study on HRQOL and Cost-effectiveness Analysis in Management of Patients With <2cm Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UW 14-500
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Thyroid Nodules
Keywords: FNAC; Small Incidental Thyroid Nodules
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FNAC (Other): patients will then be randomized routine FNAC strategy
  Interventions: Other: Fine Needle Aspiration Cytology
- No FNAC (No Intervention): patients will be randomized to watchful observation strategy (no FNAC)

INTERVENTIONS:
Other: Fine Needle Aspiration Cytology
  Other Names: FNAC
  Arms: FNAC

SUMMARY:
Ideally randomized controlled trials should be carried out to compare the cost-effectiveness between FNAC and watchful waiting but such studies are very difficult to conduct in practice because they require following up very large number of subjects for a long period of time.

The aims are to determine the health-related quality of life (HRQOL) and HRQOL preference (utility) of patients undergoing watchful observation (no FNAC) and routine FNAC, and to determine the cost-effectiveness of two strategies in managing small incidental thyroid nodules for the Chinese population in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or above
* Have life expectancy of at least 6 months
* Have an incidental nodule which measures between 1.0 to 2.0cm in the largest dimension on ultrasound guidance (USG) and has benign ultrasonographic features such as spongiform or honeycomb appearance, purely-cystic, egg shell type calcification, iso-echoic or hyper-echoic in relation to the rest of the thyroid tissue and peripheral vascularity on Doppler USG. For subjects with more than one nodule on USG, provided that the other nodules are not >2.0cm or have suspicious features (see below), they will still be eligible.
* Normal thyroid function (both serum thyroid-stimulating hormone (TSH) and free T4 levels within normal range)
* Given consent to take part in the study

Exclusion Criteria:

* Have suspicious ultrasonographic features such as microcalcifications, marked hypoechogenicity, irregular margins and / or taller than wide and intranodular vascularity on transverse view on Doppler USG that warrant a FNAC
* Nodule size > 2.0cm
* Insisting or refusing FNAC or surgical intervention despite medical reassurance
* Inability to understand or communicate in Cantonese or Chinese
* Significant cognitive impairment judged by the doctor to be unable to answer the questionnaire
* Too ill to carry out interview
* Refusal to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The measurement of HRQoL by SF-6D Health Survey | Two years
  Health-related Quality of Life (HRQoL) preference value measured by The Chinese (HK) SF-6D Health Survey will be calculated by the Hong Kong population specific algorithm. It ranges from 0 (dead) to 1 (perfect health)

SECONDARY OUTCOMES:
The effectiveness of managing small incidental thyroid nodules and treatment effect on the HRQOL of patients with thyroid carcinoma | Two years
  The effectiveness of managing small incidental thyroid nodules is quantified by quality-adjusted life years (QALYs), which will be calculated as the product of average duration of each stage (including no illness) and the SF-6D preference value for that particular health state.
  The direct health care costs of different strategies in managing small incidental thyroid nodules will be estimated using the costs published by the Government Gazette and previous literatures.
  HRQOL measured by the Chinese (Hong Kong) Short Form-12 (SF-12) Health Survey version 2 and FACT-G will be evaluated to identify these major problem of life.
  Health service utilizations of patients with thyroid neoplasm will be surveyed.
  Treatment effect on the HRQOL of patients with thyroid carcinoma will be explored.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Reiners C, Wegscheider K, Schicha H, Theissen P, Vaupel R, Wrbitzky R, Schumm-Draeger PM. Prevalence of thyroid disorders in the working population of Germany: ultrasonography screening in 96,278 unselected employees. Thyroid. 2004 Nov;14(11):926-32. doi: 10.1089/thy.2004.14.926. PMID 15671771
- [Background] Van den Bruel A, Francart J, Dubois C, Adam M, Vlayen J, De Schutter H, Stordeur S, Decallonne B. Regional variation in thyroid cancer incidence in Belgium is associated with variation in thyroid imaging and thyroid disease management. J Clin Endocrinol Metab. 2013 Oct;98(10):4063-71. doi: 10.1210/jc.2013-1705. Epub 2013 Aug 21. PMID 23966243
- [Background] Mazzaferri EL. Management of a solitary thyroid nodule. N Engl J Med. 1993 Feb 25;328(8):553-9. doi: 10.1056/NEJM199302253280807. No abstract available. PMID 8426623
- [Background] Mehanna HM, Jain A, Morton RP, Watkinson J, Shaha A. Investigating the thyroid nodule. BMJ. 2009 Mar 13;338:b733. doi: 10.1136/bmj.b733. No abstract available. PMID 19286747
- [Background] McLeod DS, Sawka AM, Cooper DS. Controversies in primary treatment of low-risk papillary thyroid cancer. Lancet. 2013 Mar 23;381(9871):1046-57. doi: 10.1016/S0140-6736(12)62205-3. Epub 2013 Mar 22. PMID 23668555
- [Background] Sosa JA, Hanna JW, Robinson KA, Lanman RB. Increases in thyroid nodule fine-needle aspirations, operations, and diagnoses of thyroid cancer in the United States. Surgery. 2013 Dec;154(6):1420-6; discussion 1426-7. doi: 10.1016/j.surg.2013.07.006. Epub 2013 Oct 2. PMID 24094448
- [Background] Bonavita JA, Mayo J, Babb J, Bennett G, Oweity T, Macari M, Yee J. Pattern recognition of benign nodules at ultrasound of the thyroid: which nodules can be left alone? AJR Am J Roentgenol. 2009 Jul;193(1):207-13. doi: 10.2214/AJR.08.1820. PMID 19542415
- [Background] Ito Y, Miyauchi A, Inoue H, Fukushima M, Kihara M, Higashiyama T, Tomoda C, Takamura Y, Kobayashi K, Miya A. An observational trial for papillary thyroid microcarcinoma in Japanese patients. World J Surg. 2010 Jan;34(1):28-35. doi: 10.1007/s00268-009-0303-0. PMID 20020290
- [Background] Pacini F. Management of papillary thyroid microcarcinoma: primum non nocere! J Clin Endocrinol Metab. 2013 Apr;98(4):1391-3. doi: 10.1210/jc.2013-1634. No abstract available. PMID 23564944
- [Background] Moon WJ, Baek JH, Jung SL, Kim DW, Kim EK, Kim JY, Kwak JY, Lee JH, Lee JH, Lee YH, Na DG, Park JS, Park SW; Korean Society of Thyroid Radiology (KSThR); Korean Society of Radiology. Ultrasonography and the ultrasound-based management of thyroid nodules: consensus statement and recommendations. Korean J Radiol. 2011 Jan-Feb;12(1):1-14. doi: 10.3348/kjr.2011.12.1.1. Epub 2011 Jan 3. PMID 21228935
- [Background] American Thyroid Association (ATA) Guidelines Taskforce on Thyroid Nodules and Differentiated
- [Derived] Wong CKH, Liu X, Lang BHH. Cost-effectiveness of fine-needle aspiration cytology (FNAC) and watchful observation for incidental thyroid nodules. J Endocrinol Invest. 2020 Nov;43(11):1645-1654. doi: 10.1007/s40618-020-01254-0. Epub 2020 Apr 19. PMID 32307641
- [Derived] Wong CKH, Lang BHH. A randomized trial comparing health-related quality-of-life and utility measures between routine fine-needle aspiration cytology (FNAC) and surveillance alone in patients with thyroid incidentaloma measuring 1-2 cm. Endocrine. 2020 Feb;67(2):397-405. doi: 10.1007/s12020-019-02129-y. Epub 2019 Nov 18. PMID 31741168
- [Derived] Wong CKH, Lang BHH, Yu HMS, Lam CLK. EQ-5D-5L and SF-6D Utility Measures in Symptomatic benign Thyroid Nodules: Acceptability and Psychometric Evaluation. Patient. 2017 Aug;10(4):447-454. doi: 10.1007/s40271-017-0220-5. PMID 28224296